CLINICAL TRIAL: NCT00098124
Title: A Phase III Pivotal, Multicenter, Double-Blind, Randomized, Placebo-Controlled Study of Milnacipran for the Treatment of Fibromyalgia
Brief Title: Study of Milnacipran for the Treatment of Fibromyalgia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MLN-MD-02
Record Dates: First submitted 2004-12-03; First posted 2004-12-06 (Estimated); Last update posted 2007-12-24 (Estimated); Status verified 2007-12

CONDITIONS: Fibromyalgia
Keywords: NSRI; milnacipran; fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Milnacipran

INTERVENTIONS:
Drug: milnacipran hydrochloride

SUMMARY:
Antidepressants of all varieties represent a common form of therapy for many chronic states including fibromyalgia. The majority of antidepressants increase the levels of serotonin or norepinephrine in the central nervous system. Milnacipran is a dual norepinephrine and serotonin reuptake inhibitor and may be effective in the treatment of fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of fibromyalgia defined by 1990 American College of Rheumatology (ACR) Criteria

Exclusion Criteria:

* Psychiatric illness
* Depression
* Suicidal risk
* Substance abuse
* Pulmonary dysfunction
* Renal impairment
* Active cardiac disease
* Liver disease
* Autoimmune disease
* Cancer
* Sleep apnea
* Inflammatory bowel disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200
Dates: Start 2004-11; Study Completion 2006-12

PRIMARY OUTCOMES:
Composite responder analysis based on pain and patient global status, with or without physical function.

SECONDARY OUTCOMES:
Quality of Life
Health Assessment Questionnaire (HAQ) Disability Index
Fatigue, sleep and cognitive assessments

CONTACTS AND LOCATIONS:
Locations (77):
- United States (77):
  - Forest Investigative Site, Birmingham, Alabama
  - Forest Investigative Site, Mobile, Alabama
  - Forest Investigative Site, Montgomery, Alabama
  - Forest Investigative Site, Peoria, Arizona
  - Forest Investigative Site, Beverly Hills, California
  - Forest Investigative Site, Sacramento, California
  - Forest Investigative Site, San Diego, California
  - Forest Investigative Site, Santa Ana, California
  - Forest Investigative Site, Spring Valley, California
  - Forest Investigative Site, Torrance, California
  - Forest Investigative Site, Colorado Springs, Colorado
  - Forest Investigative Site, Danbury, Connecticut
  - Forest Investigative Site, Stamford, Connecticut
  - Forest Investigative Site, Trumball, Connecticut
  - Forest Investigative Site, Clearwater, Florida
  - Forest Investigative Site, DeLand, Florida
  - Forest Investigative Site, Delray Beach, Florida
  - Forest Investigative Site, Jacksonville, Florida
  - Forest Investigative Site, Ocala, Florida
  - Forest Investigative Site, Ormond Beach, Florida
  - Forest Investigative Site, Palm Harbor, Florida
  - Forest Investigative Site, Pembroke Pines, Florida
  - Forest Investigative Site, Port Orange, Florida
  - Forest Investigative Site, Tamarac, Florida
  - Forest Investigative Site, Decatur, Georgia
  - Forest Investigative Site, Honolulu, Hawaii
  - Forest Investigative Site, Meridian, Idaho
  - Forest Investigative Site, Chicago, Illinois
  - Forest Investigative Site, Libertyville, Illinois
  - Forest Investigative Site, Peoria, Illinois
  - Forest Investigative Site, Evansville, Indiana
  - Forest Investigative Site, Lafayette, Indiana
  - Forest Investigative Site, Wichita, Kansas
  - Forest Investigative Site, Lexington, Kentucky
  - Forest Investigative Site, Baltimore, Maryland
  - Forest Investigative Site, Columbia, Maryland
  - Forest Investigative Site, Frederick, Maryland
  - Forest Investigative Site, Newton, Massachusetts
  - Forest Investigative Site, North Dartmouth, Massachusetts
  - Forest Investigative Site, Kalamazoo, Michigan
  - Forest Investigative Site, Flowood, Mississippi
  - Forest Investigative Site, St Louis, Missouri
  - Forest Investigative Site, Missoula, Montana
  - Forest Investigative Site, Cherry Hill, New Jersey
  - Forest Investigative Site, Clementon, New Jersey
  - Forest Investigative Site, Santa Fe, New Mexico
  - Forest Investigative Site, East Syracuse, New York
  - Forest Investigative Site, Great Neck, New York
  - Forest Investigative Site, Rochester, New York
  - Forest Investigative Site, Charlotte, North Carolina
  - Forest Investigative Site, Fayetteville, North Carolina
  - Forest Investigative Site, Hickory, North Carolina
  - Forest Investigative Site, Raleigh, North Carolina
  - Forest Investigative Site, Winston-Salem, North Carolina
  - Forest Investigative Site, Bismarck, North Dakota
  - Forest Investigative Site, Marion, Ohio
  - Forest Investigative Site, Oklahoma City, Oklahoma
  - Forest Investigative Site, Bend, Oregon
  - Forest Investigative Site, Eugene, Oregon
  - Forest Investigative Site, Medford, Oregon
  - Forest Investigative Site, Portland, Oregon
  - Forest Investigative Site, Duncanville, Pennsylvania
  - Forest Investigative Site, Warwick, Rhode Island
  - Forest Investigative Site, Orangeburg, South Carolina
  - Forest Investigative Site, Bristol, Tennessee
  - Forest Investigative Site, Chattanooga, Tennessee
  - Forest Investigative Site, Memphis, Tennessee
  - Forest Investigative Site, Austin, Texas
  - Forest Investigative Site, San Antonio, Texas
  - Forest Investigative Site, Sugarland, Texas
  - Forest Investigative Site, Richmond, Virginia
  - Forest Investigative Site, Virginia Beach, Virginia
  - Forest Investigative Site, Bellingham, Washington
  - Forest Investigative Site, Everett, Washington
  - Forest Investigative Site, Seattle, Washington
  - Forest Investigative Site, Wenatchee, Washington
  - Forest Investigative Site, Racine, Wisconsin

REFERENCES:
- [Derived] Clauw DJ, Mease P, Palmer RH, Gendreau RM, Wang Y. Milnacipran for the treatment of fibromyalgia in adults: a 15-week, multicenter, randomized, double-blind, placebo-controlled, multiple-dose clinical trial. Clin Ther. 2008 Nov;30(11):1988-2004. doi: 10.1016/j.clinthera.2008.11.009. PMID 19108787